CLINICAL TRIAL: NCT04516707
Title: Evaluation of Tolerance and Efficacy Retrospective Data of XOFIGO Prescribed by AMM in Prostate Cancer
Brief Title: Evaluation of Tolerance and Efficacy Retrospective Data of XOFIGO
Acronym: XOFIGO
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: ICM-URC 2015/75
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer; Bone Metastases; Hormone-resistant Prostate Cancer
Keywords: xofigo; clinical database
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical database — The various clinicam database will be collected solely to meet the objectives of the study.
  All data collected to create the database for this project will be anonymized

SUMMARY:
Since 13 November 2013, XOFIGO has been authorised on the European zone for the treatment of patients with prostate cancer, in the phase of resistance to castration, with symptomatic bone metastases.

bone metastases frequently give rise to "bone events" that include spinal cord compressions and pathological fractures requiring surgery or external radiotherapy.

Bone metastases are an important cause of death, disability, quality of life degradation and increase the cost of treatment.

Xofigo is indicated in patients with bone metastases symptomatic of hormone-resistant prostate cancer and without known visceral metastases.

DETAILED DESCRIPTION:
Since 13 November 2013, XOFIGO has been authorised on the European zone for the treatment of patients with prostate cancer, in the phase of resistance to castration, with symptomatic bone metastases. Prostate cancer is the most common non-cutaneous cancer in men internationally, and more than 90% of patients with hormone-resistant prostate cancer will have bone metastases.

They frequently give rise to "bone events" that include spinal cord compressions and pathological fractures requiring surgery or external radiotherapy.

Bone metastases are an important cause of death, disability, quality of life degradation and increase the cost of treatment.

There is therefore a need for bone-targeting therapeutic agents that provide a benefit in terms of survival.

Xofigo is indicated in patients with bone metastases symptomatic of hormone-resistant prostate cancer and without known visceral metastases.

This treatment appears to have fewer side effects than chemotherapy (and does not call into question subsequent chemotherapy) or that the currently available metabolic bone radiotherapy as well as better pain control and survival gain than the latter do not

ELIGIBILITY:
Inclusion Criteria:

All patients who received treatment with XOFIGO in the framework of the AMM, in France since November 2013 are potentially eligible.

Exclusion Criteria:

Patients expressing a refusal to use this research data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received treatment with XOFIGO in the framework of the AMM, in France since November 2013 are potentially eligible.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Assess the epidemiological characteristics of the treated patient population | during the treatment of XOFIGO an average of 24 weeks
  clinical data collection in the medical record

SECONDARY OUTCOMES:
Assess the presence of adverse events resulting from short-term and medium-term XOFIGO treatment | during the treatment of XOFIGO an average of 24 weeks
  clinical data collection in the medical record
Assess the number of patients who were able to benefit from the complete treatment (6 cycles) | during the treatment of XOFIGO an average of 24 weeks
  clinical data collection in the medical record
Collect the causes of premature discontinuation of treatment | during the treatment of XOFIGO an average of 24 weeks
  clinical data collection in the medical record
assess the antalgic effet of treatment (number of antalgic taken and how many time) | during the treatment of XOFIGO an average of 24 weeks
  clinical data collection in the medical record
assess the overall survival | during the treatment of XOFIGO an average of 24 weeks
  clinical data collection in the medical record

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DESHAYES, MD, Study Chair — ICM Val d'Aurelle
Locations (8):
- France (8):
  - Icm Val D'Aurelle, Montpellier, Herault
  - ICO Bordeaux, Bordeaux
  - UP Clermont Ferrand, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - IPC Marseille, Marseille
  - CRLC de Nantes, Nantes
  - APHP Hopital Cochin, Paris
  - ONCOLOPE, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harrison MR, Wong TZ, Armstrong AJ, George DJ. Radium-223 chloride: a potential new treatment for castration-resistant prostate cancer patients with metastatic bone disease. Cancer Manag Res. 2013;5:1-14. doi: 10.2147/CMAR.S25537. Epub 2013 Jan 8. PMID 23326203
- [Result] Nilsson S, Strang P, Aksnes AK, Franzen L, Olivier P, Pecking A, Staffurth J, Vasanthan S, Andersson C, Bruland OS. A randomized, dose-response, multicenter phase II study of radium-223 chloride for the palliation of painful bone metastases in patients with castration-resistant prostate cancer. Eur J Cancer. 2012 Mar;48(5):678-86. doi: 10.1016/j.ejca.2011.12.023. Epub 2012 Feb 15. PMID 22341993
- [Result] Parker CC, Pascoe S, Chodacki A, O'Sullivan JM, Germa JR, O'Bryan-Tear CG, Haider T, Hoskin P. A randomized, double-blind, dose-finding, multicenter, phase 2 study of radium chloride (Ra 223) in patients with bone metastases and castration-resistant prostate cancer. Eur Urol. 2013 Feb;63(2):189-97. doi: 10.1016/j.eururo.2012.09.008. Epub 2012 Sep 13. PMID 23000088